Yelena Wu 

RAYS: Rural Youth and Adult Sun Protection Study

Version date: 12/3/24

# RAYS: Rural Youth and Adult Sun Protection Study (Coaches) Consent Cover Letter

#### **SUMMARY**

- You are being asked to take part in a research study (RAYS). Your participation in this study is completely voluntary.
- The purpose of RAYS is to improve use of sun protective behaviors among youths living in rural communities in Utah and West Virginia.
- Your participation in this study will last about 15 months and will include receiving information about sports injury prevention or related to skin cancer prevention.
- You will be asked to complete 3 questionnaires about you and your family.
- The risks associated with study participation are minimal.
- If you decide you no longer want to participate in this study, you can contact us at any point and we will not collect any more information from you.
- We cannot guarantee any direct benefits to you, however, as compensation for your participation in the study you will receive up to \$300 in gift cards for completing questionnaires and other study-related activities.

#### **BACKGROUND**

You are being asked to take part in a research study. Before you decide, it is important for you to understand why the research is being done and what it will involve. Please take time to read the following information carefully. Take time to decide whether or not to volunteer to take part in this research study.

The purpose of this study is to help prevent skin cancer. The goal of the study is to improve use of sun protective behaviors among youths living in rural communities in Utah and West Virginia. The lead investigators for this study are Dr. Yelena Wu from the University of Utah and Huntsman Cancer Institute, Dannell Boatman from West Virginia University and Dr. Kenneth Tercyak from the Lombardi Comprehensive Cancer Center at Georgetown University.

#### **STUDY PROCEDURES**

As a coach or group leader, you will receive information and training from one of our research team members. You will be asked to encourage healthy behaviors among the children in your team or group. Each league will be randomly assigned to one of two study groups. Neither you nor the researchers choose the group you will be assigned to. The training you will receive will depend on which study group your team is assigned to. We will also observe children's sun protection behaviors during your meetings, practices, or games which our study team may video record. You will be asked to fill out a survey about your experience working with us and how the program affected the children. At the conclusion of the study, you may be contacted by the research staff for a brief interview for your feedback on delivering the program. This interview will be video or audio recorded for quality assurance. Other study activities listed above may also be video or audio recorded for later analysis by the research team. You may be contacted about study activities via email, text messages, or phone calls.



Yelena Wu 

RAYS: Rural Youth and Adult Sun Protection Study

Version date: 12/3/24

#### **RISKS**

The risk or discomforts associated with participating in this study are minimal. If you feel upset from any part of this experience, you can tell the researcher, who will tell you about resources available to help. Even though we do everything we can to protect the identity and privacy of participants, there is still a risk that data could be traced back to an individual. Once data is shared, participants can still request that their data be removed from data repositories. However, some data that have been distributed for approved research use cannot be retrieved.

### **BENEFITS**

While there are no direct benefits to you for participating in this study, you may gain awareness that you are contributing to new knowledge that may benefit others in rural communities who are at risk for skin cancer in the future.

#### PERSON TO CONTACT

If there is anything that is not clear or if you would like more information, you can e-mail the research staff at <a href="mailto:rays.study@hci.utah.edu">rays.study@hci.utah.edu</a>. If you have any complaints or concerns about this study, you can contact Dr. Yelena Wu by leaving a message at (801) 585-9427. If you feel you have been harmed as result of participation, please call Dr. Yelena Wu at (801) 585-9427, who may be reached Monday through Friday, 8am-5pm.

**Institutional Review Board:** Contact the Institutional Review Board (IRB) if you have questions regarding your rights as a research participant. Also, contact the IRB if you have questions, complaints or concerns which you do not feel you can discuss with the investigator. The University of Utah IRB may be reached by phone at (801) 581-3655 or by e-mail at <a href="irb@hsc.utah.edu">irb@hsc.utah.edu</a>.

**Research Participant Advocate:** You may also contact the Research Participant Advocate (RPA) by phone at (801) 581-3803 or by email at <a href="mailto:participant.advocate@hsc.utah.edu">participant.advocate@hsc.utah.edu</a>.

## **VOLUNTARY PARTICIPATION**

If you change your mind, you can tell us anytime that you do not want to be in this study. We will not be able to collect new information about you, and you will be withdrawn from the research study. However, we can continue to use information we have already started to use in our research, as needed to maintain the integrity of the research.

## **COSTS AND COMPENSATION TO PARTICIPANTS**

There is no cost for participating in this study. You will be compensated up to \$300 for your participation in completing study surveys and the optional post-study telephone interview. You will receive \$200 for completing a coach training session with a member of our study team, \$20 for completing survey #1 (soon), \$30 for completing survey #2 at the end of the sports season, \$30 for completing survey #3 approximately one year later, and \$20 for completing the optional telephone interview. Compensation will be provided to you directly following each study activity or questionnaire that you complete. If you do not complete all of the questionnaires or the final post-study interviews, your compensation will be prorated for the activities you did complete. Compensation will come in the form of cash-equivalent gift cards that may be physical or digital; if digital, this gift card will be issued to you by email. In addition,

FOOTER FOR IRB USE ONLY Version: K0218



University of Utah
Institutional Review Board
Approved 12/10/2024
Expires 3/7/2025
IRB\_00173007

Yelena Wu 

RAYS: Rural Youth and Adult Sun Protection Study

Version date: 12/3/24

your organization may receive a \$200 donation in appreciation of your support. This monetary donation will be given after your organization has agreed to participate in the study and will not be impacted by the withdrawal of coaches or parents from the study.

#### CONFIDENTIALITY

We will share information that identifies you with our research team members at the University of Utah at Huntsman Cancer Institute, Georgetown University at Lombardi Cancer Institute, West Virginia University, the National Cancer Institute (the study sponsor), and the University of Utah Institutional Review Board (IRB), which reviews research involving people to make sure the study protects your rights. Data will only be used for the present study and will not be saved and stored for future research. We may video and/or audio record games, practices, education sessions, post-study telephone interviews or other study activities for data analysis. Recordings will be stored in a secure manner. We will do everything we can to keep your information private but we cannot guarantee this. Study information will be kept in a secured manner and electronic records will be password protected. Your data will only be used for the present study and will not be save or shared for future research.

#### **CONSENT**

I confirm I have read the information in this consent form and have had the opportunity to ask questions. By participating in the interview and questionnaires, I agree to participate in this research. I will be provided with a copy of this form for my records.

I agree to take part in this research study as you have explained in this document.

We may contact you about future research that may be of interest to you or for other matters related to this study.

We greatly appreciate you participating in our study.

